CLINICAL TRIAL: NCT00821405
Title: Study of Peritoneal/Bowel Morphology and Splanchnic Hemodynamics by Sonography, Doppler Ultrasound and Computed Tomography in CAPD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jenq-Wen Huang, National Taiwan University Hospital
Other Study IDs: 200808062R
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Peritoneum Calcification; Bowel Wall Calcification
Keywords: Number : 250~300 patients; Correlation between PET, glucose loading and peritoneal thickness/calcification
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- peritoneal dialysis: peritoneal dialysis patient lasting for more than 3 months

SUMMARY:
Use ultrasound and computed tomography to evaluate the condition of peritoneum(thickness, calcified, etc. )and correlate the relationship between the peritoneum and other clinical condition

DETAILED DESCRIPTION:
The peritoneum after long-term peritoneal dialysis is inevitably associated with fibrosis, which further compromises the efficiency of dialysis and ultrafiltration, or even worse the development of encapsulating sclerosing peritonitis (EPS) and mortality. Transabdominal ultrasonography and computed tomography has been reported in the diagnosis of EPS. Until now, it remains a critical clinical issue to early diagnose thickening of peritoneum and preventing the formation of EPS. Transabdominal ultrasonography and computed tomography are convenient and non-invasive, and has been reported to detect the thickening of peritoneum in pediatric PD patients with a history of peritonitis.

Our recent published study confirmed the utility of transabdominal ultrasonography in the evaluation of parietal peritoneum in adult PD patients. In previous work, we examined and compared eighteen adult PD patients with PD duration of more than 7 years with other eighteen adult PD patients wit PD duration of less than 1 year. Our results indicated that sonographic thickness is associated with PD peritoneal transport characteristics but not with the duration of PD. This work was just published in Nephrology, Dialysis and Transplantation in year 2008. We believe that was the earliest published ultrasonographic study in adult PD patients.

This proposed study aims to extend from previous study by increasing examinee population to include all adult PD patients as a cross sectional observational study. We will utilize previously published sonographic examination method on PD patients (both B-mode and Doppler ultrasonography). We will collect the blood, urine and peritoneal effluent sample at the same time. We hope that through this large-scale survey we can elucidate more clearly the relationship between morphology and functional/transport characteristics of the parietal peritoneum during the natural course of renal replacement therapy with peritoneal dialysis. The results will form our basis of future longitudinal serial follow-ups for the adult PD patients. Besides, for those PD patients with suspected peritonitis, we will also perform non-invasive ultrasonographic examinations and collect relevant samples on the initial days of hospitalization in order to establish an "early predicting model" of severe, medical-refractory peritonitis by using transabdominal ultrasonography.

Peritoneum and bowel wall calcifications are found frequently in EPS, and although while pre-EPS stage. This study will utilize computed tomography to detect peritoneum and bowel calcifications in PD patients. We hope to found the relationship between calcification, peritoneum function, peritonitis frequency and future possibility of EPS.

ELIGIBILITY:
Inclusion Criteria:

* peritoneal dialysis more than 3 months

Exclusion Criteria:

* 1. pregnancy 2. received CT in recent 3 months

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients received peritoenal dialysis more than 3 months
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-09 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
peritoneal thickness, calcification, PET, glucose loading | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan